CLINICAL TRIAL: NCT02270190
Title: Evaluating the Effectivenemss of Percutaneous Tibial Nerve Stimulation as a Treatment for Tenesmus in Patients With Pelvic Floor Disorders
Brief Title: PTNS as a Treatment for Tenesmus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STH18418; 152830 (Other: IRAS)
Record Dates: First submitted 2014-10-16; First posted 2014-10-21 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Pelvic Floor Disorders
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- tenesmus patients (Other): Percutaneous Tibial Nerve Stimulation (PTNS) will be applied to all patients in the study
  Interventions: Device: Percutaneous Tibial Nerve Stimulation (PTNS)

INTERVENTIONS:
Device: Percutaneous Tibial Nerve Stimulation (PTNS)

SUMMARY:
The main research question is to see if Percutaneous Tibial Nerve Stimulation (PTNS) can improve the symptom of tenesmus in patients with pelvic floor disorders. This includes those who have rectal cancer in situ or who are post-rectal cancer treatment and have Anterior Resection Syndrome.

The secondary research questions are to see if other pelvic floor symptoms and quality of life improves for this patient group and if levels of anxiety and depression improve for these patients.

DETAILED DESCRIPTION:
The aim of the study is to discover if PTNS can be used to reduce the symptoms in those patients with tenesmus due to their pelvic floor disorders. These pelvic floor disorders include rectal cancer in situ, Anterior Resection Syndrome developed after rectal-cancer treatment, or gynaecological problems. Gynaecological problems that can cause tenesmus include radiotherapy for gynaecological cancer, ovarian cysts, pelvic organ prolapse and hysterectomy.

Currently, there is a lack of treatment options available to manage patients with tenesmus and it is hoped that PTNS will provide a simple, non-invasive treatment to this wide patient group with distressing symptoms. Assessment of symptom improvement will be used by analysing the change in scores on the COREFO, e-PAQ and HADS questionnaires, which will be completed pre and post treatment. COREFO is a validated questionnaire which includes questions specifically relating to tenesmus. e-PAQ is a validated questionnaire which looks at all aspects of the pelvic floor (bowel, urinary, vaginal, sexual) along with quality of life. HADS is a validated questionnaire classifying the patient's degree of anxiety and depression as either "normal", "borderline abnormal" or "abnormal".

There have been two pilot studies looking into the effect of PTNS in improving symptoms in Anterior Resection Syndrome patients. However, full papers have not been published of this data. These two studies assessed symptom improvement using questionnaires, but they did not use COREFO, e-PAQ or HADS, or include patients who currently have rectal cancer (i.e. not Anterior Resection Syndrome patients) or gynaecological problems and have the same tenesmus symptoms. Thus this makes this research an original proposal. e-PAQ is widely used in STH to assess pelvic floor symptoms, and thus its use here enables comparison with other patient groups who also have PTNS as a treatment option.

ELIGIBILITY:
Inclusion Criteria:

* Patients that have tenesmus who are post-rectal cancer treatment and have Anterior Resection Syndrome.
* Patients that have tenesmus who have a rectal cancer.
* Patients that have tenesmus due to a gynaecological condition.

Exclusion Criteria:

* Anyone under the age of 18.
* Anyone with a pacemaker or implantable defibrillator.
* Anyone who is prone to excessive bleeding.
* Anyone who is pregnant or is planning on becoming pregnant throughout their time in the trial.
* Anyone with diabetic neuropathy, multiple sclerosis, Parkinson's disease or peripheral neuropathy.
* Inability to provide consent for the research study.
* Anatomical limitations that would prevent successful placement of needle electrode.
* Present evidence of external full thickness rectal prolapse.
* Stoma in situ.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
improve the symptom of tenesmus in patients with pelvic floor disorders | 12 weeks
  The degree of success of the PTNS treatment will be measured by comparing the results from the COREFO, e-PAQ and HADS questionnaires before and after the 12 weeks of treatment. The treatment will be deemed successful if the post-treatment score is significantly lower than the pre-treatment score.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of General Surgery, Sheffield, South Yorkshire, United Kingdom